CLINICAL TRIAL: NCT02015143
Title: A Comprehensive Assessment and Follow up Descriptive Study on Bipolar Disorder
Acronym: CAFE-BD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University (Other)
Collaborators: Capital Medical University (Other); Shanghai Mental Health Center (Other); The First Hospital of Hebei Medical University (Other); Central South University (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Xin Yu, President, Peking University
Other Study IDs: 2011(37)
Record Dates: First submitted 2013-12-03; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Bipolar Disorder; Unipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bipolar Disorder
- Unipolar Disorder

SUMMARY:
The purpose of this study was to investigate the reliability and validity of the bipolar index (BPX) to diagnosis bipolar disorder, and to verify the stability of it in identifying bipolar disorder; the secondary purpose was to understand the dynamic changes of bipolar disorder in natural status.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old；
2. Be able to understand the content of assessment and cooperate；
3. Currently patients are depressive episode, and / or manic / hypomanic episode, also can be mood stable；
4. Currently according to diagnostic criteria of the U.S Diagnostic and Statistical Manual Fourth Edition of Mental Disease (DSM-IV) of bipolar disorder (Type I, II, rapid cycling, mixed episodes)；
5. Currently according to diagnostic criteria of the U.S Diagnostic and Statistical Manual Fourth Edition of Mental Disease (DSM-IV) of depressive disorder；
6. No other mental illness or a history of physical disease，or patients with physical disease;
7. Not received modified ECT at least four weeks or more before entering the group.

Exclusion Criteria:

1. Can not understand the content of assessment and cooperate；
2. Meet the diagnosis criteria of schizophrenia and other psychotic disorders;
3. Meet the diagnosis criteria of Diagnosis of mental retardation or pervasive developmental disorder;
4. Clinically significant neurological disease or loss of consciousness more than one hour of traumatic brain injury；

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cases were selected from the Sixth Hospital of Peking University and other eight hospitals, and they must meet the diagnosis inclusion criteria of un-bipolar and bipolar disorders. The control group of non-mood disorders will be selected from heathy population who met the following inclusion criteria of healthy controls. Informed consent must be obtained.
Sampling Method: Probability Sample
Enrollment: 970 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-03 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Test-retest reliability of the scale | one year later

SECONDARY OUTCOMES:
Cronbach's α coefficient of the scale | one year later

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Institute of Mental Health, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ma Y, Gao H, Yu X, Si T, Wang G, Fang Y, Liu Z, Sun J, Yang H, Wang X, Li J, Zhang Y, Sachs G. Bipolar diagnosis in China: Evaluating diagnostic confidence using the Bipolarity Index. J Affect Disord. 2016 Sep 15;202:247-53. doi: 10.1016/j.jad.2016.05.039. Epub 2016 May 24. PMID 27286368